CLINICAL TRIAL: NCT02588014
Title: Examining the Neural Bases of Early Visual and Auditory Processing and Emotion Recognition Deficits in Schizophrenia Using Magnetoencephalography
Brief Title: The Neural Bases of Early Visual and Auditory Processing and Emotion Recognition Deficits in Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 0018-15-SHA
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Schizophrenia; Healthy
MeSH Terms: conditions — Schizophrenia | interventions — Magnetoencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Schizophrenia: Individuals with schizophrenia
  Interventions: Other: Magnetoencephalography
- Control: Neurotypical individuals
  Interventions: Other: Magnetoencephalography

INTERVENTIONS:
Other: Magnetoencephalography — Magnetoencephalography is a non-invasive technique for investigating human brain activity. It allows the measurement of ongoing brain activity on a millisecond-by-millisecond basis, and it shows where in the brain activity is produced.
  Other Names: MEG; 4D-NeuroImage

SUMMARY:
The purpose of this project is to examine potential mechanisms that may underlie early visual and auditory perception as well as visual and auditory affect perception deficits in schizophrenia and the possible connection between these processes. Given that affect perception largely involves visual and/or auditory information processing and likely relies on intact basic visual and/or auditory perceptual mechanisms, the investigators will examine affect perception deficits within the framework of the more basic visual and auditory processes. Specifically, the investigators will examine magnetophysiological correlates of vocal and visual affect discrimination, non-affective face discrimination and voice discrimination, and simple visual and auditory stimulus discrimination, using Magnetoencephalography (MEG), to identify neural mechanisms underlying perceptual deficits, as well as their contribution to affect perception deficits in schizophrenia.

DETAILED DESCRIPTION:
Patients will be recruited from Shalvata mental health center and evaluated clinically in Shalvata mental health center. The MEG scan will take place at Bar-Ilan University at the Brain Research Center. Participants will get to and from the university with one of the researchers. Patients from the closed ward will be taken from Shalvata mental health center after receiving a signed letter from a relevant staff member allowing them to leave the hospital for the purpose of the research. At the end of the experiment hospitalized patients will be returned to the hospital and non-hospitalized ones to their preferred destination.

First stage (to take place in Shalvata): After the informed consent process a clinical evaluation will be performed. The evaluation will be administered to all participants and will include: demographic details and psychiatric history questionnaire, social functioning scale, handedness questionnaire, four-factor index of social statues for socioeconomic evaluation, Ischihara Color Blindness Test, Snellen wall chart for visual evaluation, TONI-3 test for intelligence evaluation, Hebrew version of the Manchester Short Assessment of Quality of Life, Interpersonal Reaction Index for empathy evaluation, and SCID for DSM-IV. In addition, the PANSS questionnaire will be administered to schizophrenic and schizoaffective patients. Time estimation: 1-2 hours.

Second stage (to take place at Bar-Ilan University and if necessary to be divided into two separate visits): Conducting a brain scan during a battery of tasks that will test neural mechanisms underlying visual and auditory perceptual deficits, as well as their contribution to affect perception deficits in schizophrenia at different levels of the visual and auditory processing. This stage will begin with a preparation for the scan (10-20 minutes) and then the following tasks will take place: Task 1. Gratings Perception task in which participants have to detect the 5% vertical gratings. The aim of this task is to identify the neural mechanisms underlying basic visual perceptual deficits in individuals with schizophrenia by probing the M- and P-pathways using HSF and LSF in a neutral, semantically meaningless, stimuli (~3 minutes); Task 2. Basic Color Processing Task - participants will have to detect 5% of white backgrounds among 180 red, green and gray backgrounds. The aim of this task is to asses neural mechanisms underlying basic visual perception by probing the M- and P pathways using basic color stimuli (~3minutes); Task 3. Orientation Detection Task - a task designed to identify another level of visual processing complexity, in which participants are asked to detect a missing gap in a square, displaying on green, red or gray background (~2 minutes); Task 4. Oddball Task in which participants have to detect infrequent sounds and ignore frequent and novel sounds. The aim of this task is to identify the basic neural mechanisms underlying auditory perception in individuals with schizophrenia (~13 minutes); Task 5. High and low spatial frequency facial expressions perception task. In this task participants have to identify the facial expression of the target stimuli out of three possible expressions: neutral facial expression, happy facial expression and afraid facial expression. The aim of this task is to identify the neural mechanisms underlying neutral facial perception deficit as well as affect perception deficit in individuals with schizophrenia by probing the M- and P-pathways using HSF and LSF facial stimuli (~25 minutes including breaks). Task 6. Colored Face Recognition task - Face stimuli are the same as the broad band stimuli from the previous task with one difference: faces are colored and surrounded by red, green or gray colored backgrounds. Procedure is the same as in the previous task (~25 minutes including breaks); Task 7. Processing of Affective Human Voices task in which participants have to detect and identify the content of human sounds (~15 minutes). Time estimation of the second stage of the experiment is about two hours including breaks. Total time estimation of both experimental stages: Four hours.

At the end of the experiment participants will be thanked and brought back to their destination (hospitalized participants will be returned to Shalvata Hospital). Participants will receive 200 NIS for transportation and time loss. Participants that will be screened out during the evaluation stage will receive 50 NIS for transportation and time loss.

ELIGIBILITY:
Inclusion criteria for patients:

* Capable and willing to provide informed consent
* Diagnosis of schizophrenia or schizoaffective
* Right handedness
* Corrected visual acuity
* No color blindness
* Normal hearing
* IQ ≥ 70

Inclusion Criteria for controls:

* Capable and willing to provide informed consent
* Right handedness
* Corrected visual acuity
* No color blindness
* Normal hearing
* IQ ≥ 70

Exclusion Criteria for patients:

* Left handedness
* Intellectual Disability
* Impaired vision
* Impaired hearing
* Colour blindness
* History of significant head injury or neurological illness
* Current diagnosis of substance dependence
* Metallic implants
* Severe current mental instability that precludes participation in the MEG task

Exclusion Criteria for controls:

* Psychiatric history
* Intellectual Disability
* Impaired vision
* Impaired hearing
* Colour blindness
* History of significant head injury or neurological illness
* Current diagnosis of substance dependence
* Metallic implants

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals diagnosed with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Brain responses to early visual and auditory stimuli as measured by the MEG | Immediate
  Amplitudes and brain sources of early auditory and visual components as measured by the MEG

SECONDARY OUTCOMES:
Correlation between brain responses to early visual and auditory processing and brain patterns of affect perception | Immediate
Correlation between brain responses to early visual and auditory processing and social functioning and quality of life questionnaire' grades | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Bloch, MD, Principal Investigator — Shalvata Mental Health Center